CLINICAL TRIAL: NCT02370589
Title: A Phase 1, Randomized, Observer-Blinded, Dose-Ranging Study to Evaluate the Immunogenicity and Safety of an Ebola Virus (EBOV) Glycoprotein (GP) Nanoparticle Vaccine, With or Without Matrix-M™ Adjuvant, in Healthy Subjects ≥18 to <50 Years of Age
Brief Title: Study to Evaluate the Immunogenicity and Safety of an Ebola Virus (EBOV) Glycoprotein (GP) Vaccine in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EBOV-H-101
Record Dates: First submitted 2015-02-10; First posted 2015-02-25 (Estimated); Last update posted 2021-11-24 (Actual); Status verified 2016-09

CONDITIONS: Ebola
Keywords: Ebola
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (13):
- Group A (Experimental): Day 0: Base Dose EBOV GP Vaccine; IM Day 21: Base Dose EBOV GP Vaccine; IM
  Interventions: Biological: Base Dose EBOV GP Vaccine
- Group B (Experimental): Day 0: Base Dose EBOV GP Vaccine and Matrix-M Adjuvant; IM Day 21: Base Dose EBOV GP Vaccine and Matrix-M Adjuvant; IM
  Interventions: Biological: Base Dose EBOV GP Vaccine; Biological: Matrix-M Adjuvant
- Group C (Experimental): Day 0: Base Dose EBOV GP Vaccine and Matrix-M Adjuvant; IM Day 21: Placebo; IM
  Interventions: Biological: Base Dose EBOV GP Vaccine; Biological: Placebo; Biological: Matrix-M Adjuvant
- Group D (Experimental): Day 0: 2x Base Dose EBOV GP Vaccine; IM Day 21: 2x Base Dose EBOV GP Vaccine; IM
  Interventions: Biological: 2x Base Dose EBOV GP Vaccine
- Group E (Experimental): Day 0: 2x Base Dose EBOV GP Vaccine and Matrix-M Adjuvant; IM Day 21: 2x Base Dose EBOV GP Vaccine and Matrix-M Adjuvant; IM
  Interventions: Biological: 2x Base Dose EBOV GP Vaccine; Biological: Matrix-M Adjuvant
- Group F (Experimental): Day 0: 2x Base Dose EBOV GP Vaccine and Matrix-M Adjuvant; IM Day 21: Placebo; IM
  Interventions: Biological: 2x Base Dose EBOV GP Vaccine; Biological: Placebo; Biological: Matrix-M Adjuvant
- Group G (Experimental): Day 0: 4x Base Dose EBOV GP Vaccine; IM Day 21: 4x Base Dose EBOV GP Vaccine; IM
  Interventions: Biological: 4x Base Dose EBOV GP Vaccine
- Group H (Experimental): Day 0: 4x Base Dose EBOV GP Vaccine and Matrix-M Adjuvant; IM Day 21: 4x Base Dose EBOV GP Vaccine and Matrix-M Adjuvant; IM
  Interventions: Biological: 4x Base Dose EBOV GP Vaccine; Biological: Matrix-M Adjuvant
- Group J (Experimental): Day 0: 4x Base Dose EBOV GP Vaccine and Matrix-M Adjuvant; IM Day 21: Placebo; IM
  Interventions: Biological: 4x Base Dose EBOV GP Vaccine; Biological: Placebo; Biological: Matrix-M Adjuvant
- Group K (Experimental): Day 0: 8x Base Dose EBOV GP Vaccine; IM Day 21: 8x Base Dose EBOV GP Vaccine; IM
  Interventions: Biological: 8x Base Dose EBOV GP Vaccine
- Group L (Experimental): Day 0: 8x Base Dose EBOV GP Vaccine and Matrix-M Adjuvant; IM Day 21: 8x Base Dose EBOV GP Vaccine and Matrix-M Adjuvant; IM
  Interventions: Biological: 8x Base Dose EBOV GP Vaccine; Biological: Matrix-M Adjuvant
- Group M (Experimental): Day 0: 8x Base Dose EBOV GP Vaccine and Matrix-M Adjuvant; IM Day 21: Placebo; IM
  Interventions: Biological: 8x Base Dose EBOV GP Vaccine; Biological: Placebo; Biological: Matrix-M Adjuvant
- Group N (Placebo Comparator): Day 0: Placebo; IM Day 21: Placebo; IM
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Base Dose EBOV GP Vaccine
  Arms: Group A; Group B; Group C
Biological: 2x Base Dose EBOV GP Vaccine
  Arms: Group D; Group E; Group F
Biological: 4x Base Dose EBOV GP Vaccine
  Arms: Group G; Group H; Group J
Biological: 8x Base Dose EBOV GP Vaccine
  Arms: Group K; Group L; Group M
Biological: Placebo
  Arms: Group C; Group F; Group J; Group M; Group N
Biological: Matrix-M Adjuvant
  Arms: Group B; Group C; Group E; Group F; Group H; Group J; Group L; Group M

SUMMARY:
This is a randomized, observer-blind, placebo-controlled trial in male and female subjects ≥18 to <50 years of age. Subjects will be healthy adults based on history, physical examination, and baseline clinical laboratory testing.

Approximately 230 eligible subjects will be enrolled into 1 of 13 treatment groups.

Treatments will comprise two IM doses at a 21-day interval (Day 0 and Day 21), in alternate deltoids with the test article assigned (i.e., saline placebo, dose of EBOV GP vaccine with or without Matrix-M adjuvant), in a 0.5mL injection volume.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or females, ≥18 years of age, with an upper limitation of <50 years.
2. Willing and able to give informed consent prior to study enrollment,
3. Able to comply with study requirements, and
4. Women of childbearing potential must have a negative urine pregnancy test prior to each vaccination, and will be advised through the Informed Consent process to avoid becoming pregnant over the duration of the study, and must assert that they will employ an effective form of birth control for the duration of the study. Acceptable forms of birth control are: credible history of continuous abstinence from heterosexual activity or prior surgical sterilization, hormonal contraceptives (oral, injectable, implant, patch, ring), barrier contraceptives (condom or diaphragm), and intrauterine device (IUD). Women with an adequately documented history of surgical sterility are exempt from urine pregnancy testing.

Exclusion Criteria:

1. Any ongoing, symptomatic acute or chronic illness requiring medical or surgical care.

   * Asymptomatic conditions or findings (e.g. mild hypertension, dyslipidemia) that are not associated with evidence of end-organ damage are not exclusionary provided that they are being appropriately managed and are clinically stable (i.e., unlikely to result in symptomatic illness within the time-course of this study) in the opinion of the investigator.
   * Note that illnesses or conditions may be exclusionary, even if otherwise stable, due to therapies used to treat them (see exclusion criteria 2, 5, 7, 8, 9).
2. Participation in research involving investigational product (drug/biologic/device) within 45 days before planned date of first vaccination.
3. History of a serious reaction to prior vaccination.
4. Any occupational or other exposure to Ebolaviruses or recovery from past Ebolavirus disease.
5. Received any vaccine in the 4 weeks preceding the study vaccination; or any Ebolavirus vaccine at any time.
6. Any known or suspected immunosuppressive condition, acquired or congenital, as determined by history and/or physical examination.
7. Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccine. An immunosuppressive dose of glucocorticoid will be defined as a systemic dose ≥10 mg of prednisone per day or equivalent. The use of topical and nasal glucocorticoids will be permitted. Inhaled glucocorticoids ≥500µg per day of beclamethasone or fluticasone, or 800μg per day of budesonide are exclusionary.
8. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or during the study.
9. Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature >38.0°C on the planned day of vaccine administration).
10. Known disturbance of coagulation. The use of ≤325mg of aspirin per day as prophylaxis is permitted, but use of other platelet aggregation inhibitors, thrombin inhibitors, factor Xa inhibitors, or warfarin derivatives is exclusionary, regardless of bleeding history, because these imply treatment or prophylaxis of known cardiac or vascular disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 230 (Actual)
Dates: Start 2015-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Assessment of Adverse Events, SAEs, Medically Attended Events and Significant New Medical Conditions. | Day 0 to Day 385
  Numbers and percentages (with 95% confidence intervals [CIs]) of subjects with solicited local and systemic AEs over the 7 days post-injection; and all AEs, solicited and unsolicited, including adverse changes in clinical laboratory parameters, over 84 days post-first injection. In addition, MAEs, SAEs, and SNMCs will be collected for one year after the second dose.
Immunogenicity as assessed by serum IgG antibody levels specific for EBOV Gp antigen as detected by ELISA. | Day 0 to Day 385
  * Geometric mean titer (GMT)
  * Geometric mean ratio (GMR)
  * Seroconversion rate (SCR)
  * Seroresponse rate (SRR)

SECONDARY OUTCOMES:
Immunogenicity as assessed by epitope-specific immune responses to the EBOV GP antigen measured by serum titers in a competition ELISA assay using known-neutralizing monoclonal antibodies. | Day 0 to Day 385
  * Geometric mean titer (GMT)
  * Geometric mean ratio (GMR)
  * Seroconversion rate (SCR)
  * Seroresponse rate (SRR)
Immunogenicity as assessed by serum EBOV neutralizing antibody reciprocal titers as detected by a VSV pseudotype-based method. | Day 0 to Day 385
  * Geometric mean titer (GMT)
  * Geometric mean ratio (GMR)
  * Seroconversion rate (SCR)
  * Seroresponse rate (SRR)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax, Inc.
Locations (3):
- Australia (3):
  - Q-Pharm Pty Ltd., Brisbane, Queensland
  - Nucleus Network, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia

REFERENCES:
- See also: Novavax, Inc. — http://novavax.com